CLINICAL TRIAL: NCT00066196
Title: A Phase II, Randomized, Open-Label Study Evaluating The Antitumor Activity Of MEDI-522, A Humanized Monoclonal Antibody Directed Against The Human Alpha V Beta 3 Integrin, ± Dacarbazine In Patients With Metastatic Melanoma
Brief Title: Evaluating The Antitumor Activity Of MEDI-522 With Or Without Dacarbazine In Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Luz Hammershaimb, M.D., V.P., Clinical Dev., MedImmune Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP095; NCT00081081 (obsolete NCT alias)
Record Dates: First submitted 2003-08-05; First posted 2003-08-07 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Melanoma; Malignant Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — etaracizumab; Integrins; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): Integrin + Dacarbazine
  Interventions: Biological: Integrin + Dacarbazine
- 1 (Active Comparator): MEDI-522
  Interventions: Biological: MEDI--522

INTERVENTIONS:
Biological: MEDI--522 — IV administration supplied in 10 mL vials containing 100 mg of MEDI-522 at a concentration of 10 mg/mL.
  Arms: 1
Biological: Integrin + Dacarbazine — supplied in other formulations
  Arms: 2

SUMMARY:
The primary objectives of this study are:

* To explore the antitumor activity of MEDI-522 ± DTIC in patients with metastatic melanoma.
* To determine the safety of MEDI-522 ± DTIC in this patient population.

DETAILED DESCRIPTION:
This is a Phase II, randomized, open-label, two-arm, multicenter study of MEDI 522 ± DTIC in previously untreated (other than adjuvant immunotherapy) patients with Stage IV metastatic melanoma (AJCC staging).

ELIGIBILITY:
Inclusion

Patients must meet all of the following criteria at the time of randomization:

* Histologically confirmed, unresectable, Stage IV metastatic melanoma (AJCC staging), with at least one measurable lesion defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ³ 20 mm with conventional techniques or as ³ 10 mm with spiral computed tomography (CT) scan;
* Adult men and women of at least 18 years of age at the time of randomization;
* Women of reproductive potential (defined as being <1 year post-menopausal) must have a negative serum β human chorionic gonadotropin (βhCG) pregnancy test within 3 days prior to randomization; and men and women of reproductive potential must agree to practice an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device (IUD), condom, diaphragm with spermicide, cervical cap, abstinence, or sterile sexual partner) at the time the informed consent is signed, and must agree to continue using such precautions while receiving MEDI-522 and for 30 days after the final dose of MEDI-522;
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1;
* Life expectancy of at least 16 weeks;
* WBC ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelet count ≥ 100,000/mm3;
* Bilirubin ≤ 1.5 mg/dL, aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 3 times upper limit of normal (ULN), serum creatinine ≤ 1.5 mg/dL, alkaline phosphatase ≤ 3.0 times ULN and prothrombin time (PT)/partial thromboplastin time (PTT) or international normalized ratio (INR) within normal range;
* Patients who have had prior treatment with adjuvant immunotherapy are eligible for study randomization provided that therapy ended at least 4 weeks prior to randomization;
* Patients who had prior surgery are eligible if at least 4 weeks have passed since their surgery;
* All toxicities related to prior adjuvant therapy must have resolved and all surgical wounds must have healed;
* Written informed consent and HIPAA authorization obtained from the patient prior to receipt of any study medication or beginning study procedures.

Exclusion

Patients must have none of the following at the time of randomization:

* Pregnancy or nursing;
* Prior therapy for metastatic melanoma including chemotherapy, radiotherapy, hormonal therapy, or biologics;
* Any concurrent chemotherapy, radiotherapy, immunotherapy, biologic or hormonal therapy for treatment of cancer;
* Current or planned participation (from the day of randomization through 30 days after the last dose of MEDI-522) in a research protocol in which an investigational agent or therapy may be administered;
* Received an investigational agent within 4 weeks prior to randomization;
* Known brain metastases or primary brain tumors, ocular melanoma, symptomatic pleural effusion or ascites requiring paracentesis;
* History of prior malignancies within the past 5 years other than non-melanomatous skin cancers that have been controlled, carcinoma in situ of the cervix, T1a or b prostate cancer noted incidentally during a transurethral resection of prostate (TURP) with prostate-specific antigen (PSA) values within normal limits since TURP, or superficial bladder cancer;
* History of pulmonary embolus.
* Any history or evidence of pulmonary embolism or thrombophlebitis (including deep vein thrombosis) requiring anticoagulant therapy (i.e., warfarin or heparin).
* Currently requiring therapeutic anticoagulation.
* Any evidence of hematemesis, melena, hematochezia, or gross hematuria;
* History or presence of bleeding diatheses;
* Elective surgery planned during the study period through 30 days after the last dose of MEDI-522.
* History of hypersensitivity to a previously administered monoclonal antibody.
* History of hypersensitivity to DTIC;
* History of immunodeficiency;
* Known human immunodeficiency virus (HIV) or known active viral hepatic infections;
* A prior myocardial infarction or angina, or uncontrolled/refractory hypertension within 6 months prior to randomization;
* A prior stroke or transient ischemic attack within the past 6 months;
* An active infection requiring systemic antiinfective therapy;
* Prior treatment with MEDI-522 or MEDI-523;
* A general medical or psychological condition or behavior, including substance dependence or abuse that, in the opinion of the investigator, might not permit the patient to complete the study or sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2003-08; Primary Completion 2007-04 (Estimated); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Explore antitumor activity of MEDI-522 in patients with metastatic melanoma. | Screening and after every 2 cycles of treatment until disease progression. At least 4 weeks after a patient demonstrates response.

SECONDARY OUTCOMES:
Determine the safety of MEDI-522 and/or DTIC in this patient population. | Every week until disease progression, and 30 days after disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Luz Hammershaimb, M.D., Study Director — MedImmune LLC
Locations (25):
- United States (25):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - Saint Francis Memorial Hospital, San Francisco, California
  - Cancer Institute Medical Group, Santa Monica, California
  - Medical Group of North County, Vista, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Indiana Oncology Hematology Consultants, Indianapolis, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Johns Hopkins University - SKCC at Johns Hopkins, Lutherville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Kansas City Oncology & Hematology Group, Kansas City, Missouri
  - The Melanoma Center of St. Louis, St Louis, Missouri
  - HemOnc Care, P.C., Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Discovery Alliance, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas